CLINICAL TRIAL: NCT04945239
Title: Novel Behavioral Intervention to Target Social Reward Sensitivity and Attachment
Brief Title: Amplification of Positivity to Enhance Social Connections in Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Charles Taylor, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33MH113769 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-06-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amplification of Positivity Training (6 Sessions) (Experimental)
  Interventions: Behavioral: Amplification of Positivity Training (6 Sessions)
- Stress Management Training (6 Sessions) (Active Comparator)
  Interventions: Behavioral: Stress Management Training (6 Sessions)

INTERVENTIONS:
Behavioral: Amplification of Positivity Training (6 Sessions) — 6 one-hour, clinician-administered treatment sessions focused on presenting rationale and instructions for completing positive activity exercises (e.g., gratitude, acts of kindness) designed to increase positive emotions, cognitions, and behaviors.
  Arms: Amplification of Positivity Training (6 Sessions)
Behavioral: Stress Management Training (6 Sessions) — 6 one-hour, clinician-administered treatment sessions focused on presenting rationale and instructions for activity exercises designed to decrease stress.
  Arms: Stress Management Training (6 Sessions)

SUMMARY:
The overall goal of this project is to develop a novel transdiagnostic behavioral treatment -- Amplification of Positivity (AMP) -- intended to enhance positive social connections in individuals with elevated anxiety and/or depression. Social relationship impairments are common and debilitating consequences of anxiety and depression. Existing treatments have some beneficial impact on social functioning; however, many people continue to have few and/or poor quality relationships following treatment, even after experiencing symptom relief. This study will evaluate the effects of AMP on the brain systems that have been shown to be important for establishing positive connections with others. Approximately 100 individuals (ages 18-55) seeking treatment for anxiety or depression will participate in this study. Participants will be randomly assigned with equal probability to either AMP or stress management training (SMT) (6 sessions each). Participants will be assessed at baseline and post-treatment and compared on measures assessing brain responses to social reward (primary outcome), as well as physiological, behavioral, and emotional responses to social reward (secondary outcomes). It is hypothesized that the AMP group will experience greater increases from pre- to post-treatment in activity in brain systems that regulate the processing of social reward cues (e.g., striatum) relative to participants in the SMT group. It is also hypothesized that changes in brain activation to social reward from pre- to post-treatment will be correlated with the degree of improvement in social connectedness.

ELIGIBILITY:
Inclusion Criteria:

1. Score on the Patient Health Questionnaire (PHQ)-9 is 10 or higher and/or score on the Overall Anxiety Severity and Impairment Scale (OASIS) is 8 or higher.
2. Social Connectedness Scale Revised (SCSR) < 90
3. Sheehan Disability Scale (SDS) - Social Domain ≥ 5
4. Between the ages of 18-55, inclusive.
5. Have signed informed consent document(s) indicating that the participant understands the purpose of and procedures required for the study and is willing to participate in the study.
6. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. No telephone or easy access to telephone.
2. Any substance use disorder in the past 6 months except subjects with mild alcohol, nicotine, caffeine, and marijuana use disorders will be permitted in the study, and given referrals for substance use treatment which may occur concurrently.
3. Bipolar I or Psychotic disorders.
4. Moderate to severe traumatic brain injury with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study.
5. Current and regular use (more days than not during the past 30 days) of a medication that could affect brain functioning, such as anxiolytics, antipsychotics, antidepressants, mood stabilizers, beta-blockers, sleep medications, opioids/codeine, migraine medications.
6. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos with metal dyes, unwillingness to remove body piercings, and pregnancy.
7. Non-correctable vision or hearing problems, as some tests require intact sensory functioning.
8. Concurrent psychosocial treatment: Participants completing ongoing empirically supported treatments, e.g., Cognitive behavioral therapy (CBT) targeting the presenting problem will be required to meet 12-week stability criteria so that symptom changes as a result of other psychosocial treatments are not confounded with changes due to the research.
9. Inability to complete the initial assessment battery or treatment sessions.
10. Clinical conditions assessed by the interviewer that necessitate more imminent clinical care (e.g., active suicidal ideation): These criteria are in place so participants with these other, more several symptoms can be referred for appropriate mental health services.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neural activation during social reward processing | Baseline, 10 weeks
  Change from pre- to post-assessment in neural activation in the striatum measured using functional magnetic resonance imaging (fMRI) during reward anticipation trials of the social incentive delay (SID) task. This is the primary target engagement outcome.
Change from baseline in social functioning as measured by the NIH Toolbox Companionship (Friendship and Loneliness) Surveys | Baseline, 10 weeks
  Composite score of the NIH Toolbox Friendship and Loneliness surveys. Items are answered on a 5 point scale, 1 (Never) to 5 (Always). The NIH Toolbox Friendship survey ranges from 8-40 and higher scores indicate greater perceived availability of friends or companions with whom to interact or affiliate. The NIH Toolbox Loneliness survey ranges from 5-25 and higher scores indicate greater social isolation and feelings of loneliness. The composite score will be the average of the standardized scores on the Friendship and Loneliness surveys. The composite index is the primary clinical outcome.

SECONDARY OUTCOMES:
Change from baseline in positive affect in response to a social interaction task | Baseline, 10 weeks
  The state version of the Positive and Negative Affect Schedule (PANAS) will be used to measure current ("right now") positive affect in anticipation of and following the social affiliation task. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The positive affect scale ranges from 10-50; higher scores indicate greater levels of positive affect.
Change from baseline in positive facial expressions in response to a social interaction task | Baseline, 10 weeks
  Production of positive facial expressions will be coded offline using the Computer Expression Recognition Toolbox (CERT), software that objectively codes action units (AUs) according to the Facial Action Coding System (FACS). AU12 (zygomatic major) reflects positive emotional expressions. Intensity of positive expressions will be measured by the average of AU12 values greater than zero, which identifies when an action unit is more likely to be present than absent.
Change from baseline in social approach behavior in response to a social interaction task | Baseline, 10 weeks
  Observers will rate participant behavior on self-disclosure (the degree of personal information, thoughts, and feelings revealed) and responsiveness (verbal and nonverbal displays reflecting understanding, engagement, and validation). Items are answered on a 7 point scale, 1 (not at all) to 7(very much) with higher scores indicating greater levels of social approach behavior.
Change from baseline in future approach motivation in response to a social interaction task | Baseline, 10 weeks
  The Desire for Future Interaction Scale (DFI) measures the degree to which respondents would be willing to affiliate with their conversation partner again. Items are answered on a 7 point scale, 1 (not at all) to 7 (very much) with higher scores indicating higher levels of future approach motivation.
Change from baseline in respiratory sinus arrhythmia (RSA) in response to a social interaction task | Baseline, 10 weeks
  RSA will be obtained during a resting baseline and throughout the social interaction task using the MP150 data acquisition and analysis systems. RSA is an index of parasympathetic activation and will be computed from the R-wave to R-wave interbeat interval series in the frequency range of spontaneous breathing. Higher levels of RSA indicate higher levels of parasympathetic activation. RSA reactivity will be computed by subtracting RSA during baseline from RSA during the social interaction.

OTHER OUTCOMES:
Change from baseline in social functioning as measured by the NIH Toolbox Friendship Survey | Baseline, 10 weeks
  NIH Toolbox Friendship survey. Items are answered on a 5 point scale, 1 (Never) to 5 (Always). The NIH Toolbox Friendship survey ranges from 8-40 and higher scores indicate greater perceived availability of friends or companions with whom to interact or affiliate.
Change from baseline in social functioning as measured by the NIH Toolbox Loneliness Survey | Baseline, 10 weeks
  NIH Toolbox Loneliness survey. Items are answered on a 5 point scale, 1 (Never) to 5 (Always). The NIH Toolbox Loneliness survey ranges from 5-25 and higher scores indicate greater social isolation and feelings of loneliness.
Change from baseline in social functioning as measured by the Social Network Survey | Baseline, 10 weeks
  The Social Network Survey measures social functioning by looking at the size and density of a participants social network. Higher scores indicate larger social networks.
Change from baseline in social connectedness as measured by the Social Connectedness Scale Revised (SCSR) | Baseline, 10 weeks
  The SCSR measures social connectedness. Items are answered on a 6 point scale, 1 (Strongly disagree) to 6 (Strongly agree). The SCSR ranges from 20-120 and higher scores indicate greater levels of social connectedness.
Change from baseline in functional impairment as measured by the Sheehan Disability Scale | Baseline, 10 weeks
  The Sheehan Disability Scale measures functional impairment. Items are rated on a 11 point scale, 0 (Not at all) to 10 (Extremely). The scale ranges from 0-30 and higher scores indicate higher levels of functional impairment.
Change from baseline in positive affect as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect - Short Form 15a survey | Baseline, 10 weeks
  The PROMIS Positive Affect - Short Form 15a survey measures positive affect. Items are answered in a 5 point scale, 1 (Not at all) to 5 (Very much). The PROMIS Positive Affect - Short Form 15a survey ranges from 15-75 and higher scores indicate higher levels of positive affect.
Change from baseline in positive affect as measured by Positive and Negative Affect Schedule | Baseline, 10 weeks
  The Positive and Negative Affect Schedule (PANAS) measures positive affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The positive affect scale ranges from 10-50 and higher scores indicate greater levels of positive affect.
Change from baseline in positive affect as measured by Modified Differential Emotions Scale | Baseline, 10 weeks
  The Modified Differential Emotions Scale (mDES) measures positive emotions. Items are answered on a 5 point scale, 0 (Never/Not at all) to 4 (Most of the time/Extremely). Higher scores on the positive emotions sub-scale indicate higher levels of positive emotion.
Change from baseline in psychological well-being as measured by PROMIS General Life Satisfaction - Short Form 5a survey | Baseline, 10 weeks
  The PROMIS General Life Satisfaction - Short Form 5a survey measures psychological well-being. The PROMIS General Life Satisfaction items are answered on a 7 point scale, 1 (Strongly disagree) to 7 (Strongly agree). The PROMIS General Life Satisfaction survey ranges from 5-25 and higher scores indicate higher levels of life satisfaction.
Change from baseline in psychological well-being as measured by PROMIS Meaning and Purpose - Short Form 6a survey | Baseline, 10 weeks
  The PROMIS Meaning and Purpose - Short Form 6a survey measure psychological well-being. The PROMIS Meaning and Purpose items are answered on a 5 point scale, 1 (Not at all) to 5 (Very much). The PROMIS Meaning and Purpose survey ranges from 6-30 and higher scores indicate higher levels of self reported meaning and purpose in ones life.
Change from baseline in negative affect as measured by the Positive and Negative Affect Schedule | Baseline, 10 weeks
  The Positive and Negative Affect Schedule (PANAS) measures negative affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The negative affect scale ranges from 10-50 and lower scores indicate lower levels of negative affect.
Change from baseline in anxiety as measured by PROMIS Anxiety 7a survey | Baseline, 10 weeks
  The PROMIS Anxiety 7a survey measures symptoms of anxiety. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 7-35 and higher scores indicate higher levels of anxiety.
Change from baseline in depression as measured by PROMIS Depression 8b survey | Baseline, 10 weeks
  The PROMIS Depression 8b survey measures symptoms of depression. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 8-45 and higher scores indicate higher levels of depression.
Change from baseline in perceived emotional support as measured by the NIH Toolbox Emotional Support | Baseline, 10 weeks
  The NIH Toolbox Emotional Support measures perceived emotional support from others. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 8-40 and higher scores indicate greater perceived emotional support.
Change from baseline in social activity satisfaction as measured by the PROMIS Satisfaction with Participation in Discretionary Social Activities - Short Form 7a | Baseline, 10 weeks
  The PROMIS Satisfaction with Participation in Discretionary Social Activities measures perceived satisfaction with one's discretionary social activities such as leisure activity and relationships with friends. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 7-35 and higher scores indicate greater perceived emotional support.
Change from baseline in social activity satisfaction as measured by the PROMIS Satisfaction with Social Roles and Activities | Baseline, 10 weeks
  The PROMIS Satisfaction with Social Roles and Activities measures perceived satisfaction with one's social roles such as work and family responsibilities. Items are rated on a 5 point scale, 1 (Never) to 5 (Always). The scale ranges from 8-40 and higher scores indicate greater satisfaction with social roles.
Change from baseline in social anxiety symptoms as measured by the Liebowitz Social Anxiety Scale (LSAS) | Baseline, 10 weeks
  The LSAS measures level of fear/anxiety and avoidance of social situations. Items are rated on a 4 point scale, 0 (None/Never) to 3 (Severe/Usually). The Fear subscale and the Avoidance subscale both range from 0-72 (total LSAS score range 0-144), with higher scores indicating greater fear and avoidance of social situations.
Change from baseline in social anhedonia as measured by the Specific Loss of Interest and Pleasure Scale (SLIPS) | Baseline, 10 weeks
  The SLIPS measures changes in anhedonic symptoms independent of broader depressive symptoms. Items are rated on a 4 point scale, 0 to 3, representing a range of anhedonia in various social situations. The scale ranges from 0-69 and higher scores indicate higher levels of social anhedonia.
Change from baseline in anxiety-related general distress as measured by Mood and Anxiety Symptom Questionnaire - Short Form (MASQ-SF) | Baseline, 10 weeks
  The MASQ-SF measures mood and anxiety symptoms with 4 subscales. Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The General Distress Anxiety subscale ranges from 11-55 and higher scores indicate greater anxiety-related distress.
Change from baseline in depression-related general distress as measured by Mood and Anxiety Symptom Questionnaire - Short Form (MASQ-SF) | Baseline, 10 weeks
  The MASQ-SF measures mood and anxiety symptoms with 4 subscales. Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The General Distress Depression subscale ranges from 12-60 and higher scores indicate greater depression-related distress.
Change from baseline in anxious arousal as measured by Mood and Anxiety Symptom Questionnaire - Short Form (MASQ-SF) | Baseline, 10 weeks
  The MASQ-SF measures mood and anxiety symptoms with 4 subscales. Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The Anxious Arousal subscale ranges from 17-85 and higher scores indicate greater anxious arousal.
Change from baseline in anhedonic depressive symptoms as measured by Mood and Anxiety Symptom Questionnaire - Short Form (MASQ-SF) | Baseline, 10 weeks
  The MASQ-SF measures mood and anxiety symptoms with 4 subscales. Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The Anhedonic Depression subscale ranges from 22-110 and higher scores indicate higher levels of anhedonia.
Change from baseline in emotion regulation strategies as measured by Emotion Regulation Questionnaire | Baseline, 10 weeks
  The ERQ measures habitual use of the emotion regulation strategies expressive suppression and cognitive reappraisal. Items are rated on a 7 point scale, 1 (Strongly Disagree) to 7 (Strongly Agree). The Expressive Suppression subscale ranges from 1-28 and the Cognitive Reappraisal subscale ranges from 1-42, with higher scores indicating greater use of each respective emotion regulation strategy.
Change from baseline in regulation of positive emotional experiences as measured by Responses to Positive Affect Questionnaire (RPA) | Baseline, 10 weeks
  The RPA measures how individuals regulate positive emotional experiences. Items are rated on a 4 point scale, 1 (Almost never) to 4 (Almost always). The Emotion-Focused Positive Rumination subscale ranges from 5-20. The Self-Focused Positive Rumination subscale ranges from 4-16. The Dampening subscale ranges from 8-40. Higher scores on each subscale indicate greater use of each respective positive emotion regulation strategy.
Change from baseline in capacity to cope with adversity as measured by Connor-Davidson Resilience Scale (CD-RISC-10) | Baseline, 10 weeks
  The CD-RISC-10 measures an individual's capacity to cope with adversity. Items are rated on a 5 point scale, 0 (Not true at all) to 4 (True nearly all the time). The scale ranges from 0-40 and higher scores indicate greater capacity to cope with adversity.
Change from baseline in trait anxious and avoidant attachment as measured by the Experiences in Close Relationships-Revised (ECR-R) | Baseline, 10 weeks
  The ECR-R measures an individual's attachment style and experiences in close relationships. Items are rated on a 7 point scale, 1 (Disagree) to 7 (Agree). The Attachment Anxiety and the Attachment Avoidance subscales both range from 8-56, and higher scores indicate greater attachment insecurity.
Change from baseline in self-efficacy beliefs in the domain of emotion regulation as measured by the Regulatory Emotional Self-Efficacy Scale (RESE) | Baseline, 10 weeks
  The RESE measures emotion regulation self-efficacy beliefs. Items are rated on a 5 point scale, 1 (Not well at all) to 5 (Very well). The scale ranges from 1-60 and higher scores indicate greater emotion regulation self-efficacy beliefs.
Change from baseline in perceived self-efficacy as measured by the PROMIS Self-Efficacy (General; 4 item) | Baseline, 10 weeks
  The PROMIS Self-Efficacy - General measures an individual's perceived capacity to handle difficult problems and unexpected events. Items are rated on a 5 point scale, 1 (I am not at all confident) to 5 (I am very confident). The scale ranges from 4-20 and higher scores indicate greater perceived self-efficacy.
Change from baseline in trait mindfulness as measured by the Five-Facet Mindfulness Questionnaire-Short Form (FFMQ-SF) - 15 item | Baseline, 10 weeks
  The FFMQ-SF measures trait mindfulness by assessing 5 separate facets of mindfulness, including acting with awareness, observing, describing, non-judging, and non-reacting. Items are rated on a 5 point scale, 1 (Never or very rarely true) to 5 (Very often or always true). Each subscale ranges from 3-15, with higher scores indicating greater mindfulness.
Change from baseline in interpersonal difficulties based on a circumplex model of personality as measured by the Inventory of Interpersonal Problems-32 (IIP-32) | Baseline, 10 weeks
  The IIP-32 measures interpersonal difficulties with 8 subscales: Domineering/Controlling, Vindictive/Self-Centered, Cold/Distant, Socially Inhibited, Nonassertive, Overly Accommodating, Self-Sacrificing, and Intrusive/Needy. Items are rated on a 5 point scale, 0 (Not at all) to 4 (Extremely). Each subscale ranges from 0-20, and higher scores indicate greater interpersonal difficulties.
Change from baseline in low arousal positive affect experienced during the past week as measured by the Relaxed and Safe/Content Scales on the Types of Positive Affect Scale (TPAS) | Baseline, 10 weeks
  The TPAS measures levels of low arousal positive emotion, such as "calm" or "at ease" during the past week. Items are rated on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The scale ranges from 10-50 and higher scores indicate higher levels of low arousal positive emotion.
Change from baseline in mood during a social interaction task as measured by Subjective Mood Ratings | Baseline, 10 weeks
  Subjective Mood ratings measure levels of anxiety, positive and negative mood, connectedness, and emotion suppression throughout a social interaction task. Each emotion is rated with a single-item, 0 (Not at all) to 100 (Extremely). Greater scores on each subscale indicate higher levels of each respective emotion or emotion suppression.
Change from baseline in behavior during a social interaction task as measured by the Social Judgment Questionnaire (SJQ) | Baseline, 10 weeks
  The SJQ measures two dimensions of behavior: Anxiety-Related Behavior and Social Approach Behavior. Each item is rated on a 7 point scale, 1 (Not at all) to 7 (Very much). The Anxiety-Related Behavior subscale ranges from 6-42, and the Approach-Related Behavior subscale ranges from 5-35, with higher scores on each subscale indicating more anxiety- and approach-related behavior, respectively.
Change from baseline in perceived connectedness to an interaction partner during a social interaction task as measured by the Inclusion of Other in the Self (IOS) | Baseline, 10 weeks
  The IOS measures how close or interconnected the respondent feels with a conversation partner, with respondents choosing from 7 pairs of circles representing "Self" and "Other" that range from barely touching to almost completely overlapping. The single item is rated on a 7 point scale, 1 (No overlap) to 7 (most overlap), which higher scores indicating greater perceived closeness.
Change from baseline in safety behaviors during a social interaction task as measured by the Safety Behaviors Questionnaire (SBQ) | Baseline, 10 weeks
  The SBQ uses self-report to measure the use of safety behaviors intended to minimize or eliminate anticipated feared social outcomes. Items are rated on a 9 point scale, 0 (Not at all) to 8 (All the time). The scale ranges from 0-208 and higher scores indicate greater use of safety behaviors.
Change from baseline in suicidal ideation as measured by the Columbia Suicide Severity Rating Scale (CSSRS) | Baseline, 10 weeks
  The CSSRS is a measure of suicidal ideation that asks about thoughts and feelings relating to suicide since the participant's last visit. Items are rated with a binary yes/no response, and are ordered to assess suicidal ideation with increasing risk of suicidal behavior, from Item 1 (Wish to be Dead) to Item 5 (Active Suicidal Ideation with Specific Plan and Intent). The score ranges from 0-5, based on the highest item rated yes.
Change from baseline in state positive affect, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks
  The EMA state positive emotion scale measures momentary positive affect at the time of the survey prompt. Sample items include "content" and "enthusiastic." Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The scale ranges from 4-20, and higher scores indicate greater momentary positive affect.
Change from baseline in state negative affect, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks
  The EMA state negative emotion scale measures momentary negative affect at the time of the survey prompt. Sample items include "anxious/nervous" and "sluggish." Items are rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). The scale ranges from 4-20, and higher scores indicate greater momentary negative affect.
Change from baseline in perceived quality of social interactions, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks
  Perceived quality of social interactions measures the perceived acceptance, connectedness, and satisfaction during a reported social interaction. The items are rated on a 5 point scale, 1 (Not at all) to 7 (Extremely). The scale ranges from 3-21, and higher scores indicate greater perceived quality of a social interaction.
Change from baseline in perceived social connectedness/loneliness, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks
  Throughout the day, connectedness and loneliness are each measured with a single item rated on a 5 point scale, 1 (Not at all) to 5 (Extremely). During reported interactions, connectedness is measured with a single item rated on a 7 point scale, 1 (Not at all) to 7 (Extremely). At the end of the day, perceived social connectedness and loneliness are each rated with a single item rated on a 7 point scale, 1 (Not at all) to 7 (Very).
Proportion of times engaged in social interaction, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks
Number of social interactions per day, measured via Ecological Momentary Assessment | Baseline 5-day period to Post-Intervention 5-day period, 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463